CLINICAL TRIAL: NCT01526083
Title: Single-center, Open-label, Randomized 2-way Crossover Study of the Effect of Lacosamide 200 mg Twice Daily on the Single-dose Pharmacokinetics and Pharmacodynamics of Warfarin (25 mg) in Healthy Male Volunteers
Brief Title: Effect of Lacosamide 200 mg Twice a Day (Bid) on Single Dose Warfarin 25 mg in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EP0013; 2011-004911-21 (EudraCT Number)
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: Male Healthy Volunteers
MeSH Terms: interventions — Lacosamide; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single dose of Warfarin on day 3 (Other): Single dose of Warfarin on day 3 of a 7 day course of Lacosamide 200 mg BID
  Interventions: Other: Lacosamide
- Single dose of Warfarin (Other)
  Interventions: Other: Warfarin

INTERVENTIONS:
Other: Lacosamide — Strength: 200 mg, Form: Tablet, Frequency: Twice daily, Duration: 9 days
  Other Names: Vimpat
  Arms: Single dose of Warfarin on day 3
Other: Warfarin — Strength: 5 mg, Form: Tablet, Frequency: 1 single dose in each period
  In total, during the two periods, each healthy volunteer will receive 2 single doses 3 weeks apart.
  Duration: single dose
  Other Names: Coumadin
  Arms: Single dose of Warfarin

SUMMARY:
The purpose of this study is to investigate the effect of Lacosamide 200 mg twice a day (bid) on single dose pharmacokinetics (PK) and pharmacodynamics (PD) of Warfarin (25 mg) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers 18-55 years of age
* BMI 18.0-30.0 kg/m2 and weight at least 50 kg
* Tympanic body temperature 35.0-37.5°C (95 and 99.5°F) inclusive

Exclusion Criteria:

* Volunteer has participated or is participating in any other clinical studies of investigational drug or another Investigational Medicinal Product (IMP) within the last 3 months
* Volunteer is not healthy (eg, taking any drug treatments, excessive amount of alcohol, cigarettes or caffeine, having any medical or emotional/psychological problems, a drug/alcohol abuse, having abnormal safety parameters)
* Volunteer is taking Warfarin or Non Steroidal Anti-Inflammatory Drug (NSAID)
* Volunteer has history of suicide attempt
* Volunteer has history of coagulation abnormalities, occult blood in stool, gastrointestinal ulcer, surgery within 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Area under the Warfarin plasma concentration versus time curve from time 0 to infinity, AUC (Warfarin) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose in each treatment period
Area under the Warfarin plasma concentration versus time curve from time 0 to the last quantifiable level, AUC0-t(Warfarin) | Multiple sampling from 0 -168 hours following administration of a single warfarin dose in each treatment period
Maximum Warfarin plasma concentration (Cmax) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose in each treatment period
Maximum prothrombin time (PTmax) | Multiple sampling from 0 -168 hours following administration of a single warfarin dose in each treatment period
Warfarin area under the prothrombin time (PT) versus time curve (PTAUC) | Multiple sampling from 0 -168 hours following administration of a single warfarin dose in each treatment period
Warfarin maximum international normalized ratio (INRmax) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose in each treatment period
Warfarin area under the International Normalized Ratio (INR) versus time curve (INRAUC) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose in each treatment period

SECONDARY OUTCOMES:
Lacosamide trough plasma concentration (Ctrough) | Morning pre dose sample on Days 3-10 or Days 24 -30 of Lacosamide BID dosing
Time of maximum Warfarin plasma concentration (Tmax) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose
Terminal half-life of Warfarin (T ½) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose
Apparent total body clearance of Warfarin (CL /F) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose
Apparent volume of distribution of Warfarin (V /F) | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose
First order terminal elimination rate constant of Warfarin | Multiple sampling from 0 -168 hours following administration of a single Warfarin dose
CYP2C9 genotype | Single measurement on Day 1
VKORC1 genotype | Single measurement on Day 1
Occurrence of at Least One Treatment-emergent Adverse Event (TEAE) during the duration of the study | Duration of study is approximately 32 days
Change from Baseline in Pulse Rate at 4 h post dose | From pre dose to 4 h post dose Warfarin administration in each treatment period
  40-90 bpm
Change from Baseline in Pulse Rate at 12 h post dose | From pre dose to 12 h post dose Warfarin administration in each treatment period
  40-90 bpm
Change from Baseline in Pulse Rate at 24 h post dose | From pre dose to 24 h post dose Warfarin administration in each treatment period
  40-90 bpm
Change from Baseline in Pulse Rate at 4 h post dose | From pre dose to 4 h post dose Lacosamide (LCM) administration
  40-90 bpm
Change from Baseline in Pulse Rate at 12 h post dose | From pre dose to 12 h post dose LCM administration
  40-90 bpm
Change from Baseline in Systolic Blood Pressure at 4 h post dose | From pre dose to 4 h post dose Warfarin administration in each treatment period
Change from Baseline in Systolic Blood Pressure at 12 h post dose | From pre dose to 12 h post dose Warfarin administration in each treatment period
Change from Baseline in Systolic Blood Pressure at 24 h post dose | From pre dose to 24 h post dose Warfarin administration in each treatment period
Change from Baseline in Systolic Blood Pressure at 4 h post dose | From pre dose to 4 h post dose LCM administration
Change from Baseline in Systolic Blood Pressure at 12 h post dose | From pre dose to 12 h post dose LCM administration
  40-90 bpm
Change from Baseline in Diastolic Blood Pressure at 4 h post dose | From pre dose to 4 h post dose Warfarin administration in each treatment period
Change from Baseline in Diastolic Blood Pressure at 12 h post dose | From pre dose to 12 h post dose Warfarin administration in each treatment period
Change from Baseline in Diastolic Blood Pressure at 24 h post dose | From pre dose to 24 h post dose Warfarin administration in each treatment period
Change from Baseline in Diastolic Blood Pressure at 4 h post dose | From pre dose to 4 h post dose LCM administration
Change from Baseline in Diastolic Blood Pressure at 12 h post dose | From pre dose to 12 h post dose LCM administration
  40-90 bpm
Change from Baseline in Body Temperature at 4h post dose | From pre dose to 4 h post dose Warfarin administration in each treatment period
Change from Baseline in Body Temperature at 12 h post dose | From pre dose to 12 h post dose Warfarin administration in each treatment period
Change from Baseline in Body Temperature at 24 h post dose | From pre dose to 24 h post dose Warfarin administration in each treatment period
Change from Baseline in Body Temperature at 4 h post dose | From pre dose to 4 h post dose LCM administration
Change from Baseline in Body Temperature at 12 h post dose | From pre dose to 12 h post dose LCM administration
  40-90 bpm

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — 1 877 822 9493
Locations (1):
- 001, Zuidlaren, Netherlands